CLINICAL TRIAL: NCT07159490
Title: Lower Limb Prostheses for Individuals Who Carry Infants, Toddlers, and Other Loads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Glenn K. Klute, PhD, Research Career Scientist / Affiliate Professor, VA Puget Sound Health Care System
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1588093
Record Dates: First submitted 2022-06-01; First posted 2025-09-08 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Amputation; Prosthesis User
Keywords: Lower limb prosthesis; Transtibial amputation; Below knee amputation; Biomechanics
MeSH Terms: interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: This study will employ a within-subject experimental design. Each participant will wear, in randomized order, a standard-of-care prosthetic foot, this same prosthetic foot with a heel-stiffening wedge, this same prosthetic foot but one category stiffer, a dual keel prosthetic foot intended for load carriage applications, and a powered ankle-foot purported to adapt to changing loads. All study prostheses are commercially available. Each participant, wearing each of the study prostheses, will walk overground with no added load and four added load conditions of 13.6 kg: anterior, posterior, intact-side carry, and prosthetic-side carry. The load condition will be presented in block randomized order.
Who Masked: Participant
Masking Description: A sock and foot cover to blind the participants to the study prostheses when possible (use of the powered ankle-foot will be obvious).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- No added load (Experimental): Study participants will walk with no added load.
  Interventions: Device: Standard-of-care prosthetic foot; Device: Standard-of-care prosthetic foot with heel-stiffening wedge; Device: Standard-of-care prosthetic foot of one category greater stiffness; Device: Dual keel prosthetic foot; Device: Powered ankle-foot
- Anterior added load (Experimental): Study participants will walk with 13.6 kg (30 lbs) of added load on their anterior side.
  Interventions: Device: Standard-of-care prosthetic foot; Device: Standard-of-care prosthetic foot with heel-stiffening wedge; Device: Standard-of-care prosthetic foot of one category greater stiffness; Device: Dual keel prosthetic foot; Device: Powered ankle-foot
- Posterior added load (Experimental): Study participants will walk with 13.6 kg (30 lbs) of added load on their posterior side.
  Interventions: Device: Standard-of-care prosthetic foot; Device: Standard-of-care prosthetic foot with heel-stiffening wedge; Device: Standard-of-care prosthetic foot of one category greater stiffness; Device: Dual keel prosthetic foot; Device: Powered ankle-foot
- Intact-side added load (Experimental): Study participants will walk with 13.6 kg (30 lbs) of added load on their intact side.
  Interventions: Device: Standard-of-care prosthetic foot; Device: Standard-of-care prosthetic foot with heel-stiffening wedge; Device: Standard-of-care prosthetic foot of one category greater stiffness; Device: Dual keel prosthetic foot; Device: Powered ankle-foot
- Prosthetic-side added load (Experimental): Study participants will walk with 13.6 kg (30 lbs) of added load on their prosthetic side.
  Interventions: Device: Standard-of-care prosthetic foot; Device: Standard-of-care prosthetic foot with heel-stiffening wedge; Device: Standard-of-care prosthetic foot of one category greater stiffness; Device: Dual keel prosthetic foot; Device: Powered ankle-foot

INTERVENTIONS:
Device: Standard-of-care prosthetic foot — Widely prescribed prosthetic foot of stiffness category appropriate to the participant's body weight and activity level.
  Other Names: Sierra, Freedom Innovations
Device: Standard-of-care prosthetic foot with heel-stiffening wedge — Widely prescribed prosthetic foot with a wedge inserted between the heel and foot keels intended to stiffen the behavior of the heel.
  Other Names: Sierra, Freedom Innovations
Device: Standard-of-care prosthetic foot of one category greater stiffness — Widely prescribed prosthetic foot of one stiffness category greater than usually prescribed based on the participant's body weight and activity level.
  Other Names: Sierra, Freedom Innovations
Device: Dual keel prosthetic foot — A prosthetic foot with two forefoot keels intended for load carriage applications.
  Other Names: Thrive, Freedom Innovations
Device: Powered ankle-foot — A powered prosthetic ankle-foot.
  Other Names: Empower, Otto Bock

SUMMARY:
The aim of this research is to identify the prosthetic foot that results in improved walking performance when individuals with lower limb amputation carry infants, toddlers, or other loads.

DETAILED DESCRIPTION:
The natural lower limbs provide important biomechanical functions such as body weight support, forward propulsion, and balance control during ambulation. When the loads borne by the lower limbs change, lower limb muscle activation responds accordingly to enable seamless continuation of biomechanical function. These loads can change suddenly, such as when carrying an infant, toddler, or other load like a heavy backpack. For individuals with a lower limb amputation, these sudden changes to weight-bearing loads can be problematic because they can negatively impact walking performance. One reason walking performance may suffer is that the properties of most prosthetic limbs, such as their stiffness, are constant and do not change to suit varying load conditions. Another reason is that the most widely prescribed prosthetic feet do not have motors, sensors, or brain-like controllers that act to replace the neuromuscular system of the amputated limb. Regardless of the reason, no evidence exists to guide prescription practice for veterans who walk with a prosthesis and experience sudden load changes.

The aim of this research is to identify the prosthetic foot that results in improved walking performance when individuals with lower limb amputation carry infants, toddlers, or other loads. The investigators will conduct a human subject experiment with help of twenty individuals with below-knee amputations. Study participants will walk on a treadmill with no added load and four added load conditions using a weighted pack (13.6 kg or ~30 lbs) to simulate an infant, toddler, or other load. The four conditions include the pack strapped to their front, their back, and carried with their arms on the intact limb side and the prosthetic limb side. Each participant will wear a usual prosthetic foot, this same foot with a heel-stiffening wedge, the same prosthetic foot but one category stiffness higher, a new-to-market dual keel prosthetic foot intended for load carrying situations, and a powered ankle foot prosthesis. The results from these experiments will aid clinicians in specifying the best prosthesis for individuals with lower limb amputations who frequently carry infants, toddlers, or other loads.

For individuals who wear a lower limb prosthesis while carrying infants, toddlers, or other loads, this research will provide evidence to support prosthesis prescription practice that reduces undesirable compensatory responses to load carriage. The objective is to help clinicians select among currently available solutions to enable individuals with lower limb loss to achieve their life and work goals.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral transtibial amputee
2. Have been fitted with and used a prosthesis for at least six months
3. Do not use heel stiffening wedges or bumpers in their as-prescribed prosthesis
4. Wear their prosthesis for at least four hours per day
5. Are moderately active by self-report
6. Can be fitted with the study prostheses (prosthetic foot size, stiffness category and build heights)

Exclusion Criteria:

1. Do not have a proper fit and suspension and one cannot be achieved with clinical resources
2. Presence of disorder, pain, or injury other than amputation that interferes with gait

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Klute, PhD, Principal Investigator — VA Puget Sound Care System
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset in machine-readable format will be created and shared for all individual participant data (IPD) that underlie results in a publication. The investigators will follow 164.514(a) of the HIPAA Privacy Rule for de-identification of IPD.
Time Frame: Within six months after publication of final study findings.
Access Criteria: Open-source data repository (e.g., PubMed Central)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One enrolled participant decided they were no longer interested in participating after the first visit (alignment and acclimation) but before the second visit (randomization).
Groups:
- Individuals With Lower Limb Amputation: In this cross-over study, all subjects were asked to with no added load and four added load conditions using a weighted pack (13.6 kg or ~30 lbs) to simulate an infant, toddler, or other load. The four conditions include the pack strapped to their front (anterior), their back (posterior), and carried with their arms on the intact limb side and the prosthetic limb side. The load conditions were presented in block randomized order.
  While performing each of these activities, the participant wore five different prosthetic feet. These prosthetic feet included a standard-of-care prosthetic foot, this same prosthetic foot with a heel-stiffening wedge, this same prosthetic foot but one category stiffer, a dual keel prosthetic foot intended for load carriage applications, and a powered ankle-foot purported to adapt to changing loads. The prosthetic feet were worn in randomized order and the subject was blinded to the study foot using a sock and foot cover when possible (wearing a powered ankle-foot is obvious to the participant).
  The study was conducted over two visits with overnight rest in between each visit. During the first study visit, each study foot was aligned to the participant's prosthesis and wore each for at least 15 minutes. During the second study visit, the participant walked wearing each of the five different study feet while performing each of the five different load conditions.
Period: Overall Study
Arm/Group | Individuals With Lower Limb Amputation
Started | 12
**Standard-of-care prosthetic foot | 12
Walking with no added load | 12
Walking with anterior load | 12
Walking with posterior side | 12
Walking with load on prosthetic side | 12
Walking with load on intact side | 12
**Standard-of-care prosthetic foot of one category greater stiffness | 12
Walking with no added load | 12
Walking with anterior load | 12
Walking with posterior load | 12
Walking with load on prosthetic side | 12
Walking with load on intact side | 12
**Standard-of-care prosthetic foot with heel-stiffening wedge | 12
Walking with no added load | 12
Walking with anterior load | 12
Walking with posterior load | 12
Walking with load on prosthetic side | 12
Walking with load on intact side | 12
**Dual keel prosthetic foot | 12
Walking with no added load | 12
Walking with anterior load | 12
Walking with posterior load | 12
Walking with load on prosthetic side | 12
Walking with load on intact side | 12
**Powered ankle-foot | 7 (Five participants had long residual limbs and could not accommodate the build height of the powered ankle-foot.)
Walking with no added load | 7
Walking with anterior load | 7
Walking with posterior load | 7
Walking with load on prosthetic side | 7
Walking with load on intact side | 7
Completed | 7
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Individuals With Lower Limb Amputation
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 3
  Unknown or Not Reported | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Vertical Ground Reaction Force Impulse (Normalized)
Description: A measure of body support. Normalized by body mass, including the mass of the load when applicable.
Time Frame: During study visit (approximately 3 hours)
Measure: Mean (Standard Error); unit: Newtons*seconds/kg
Arm/Group | Standard-of-care Prosthetic Foot | Standard-of-care Prosthetic Foot With Heel-stiffening Wedge | Standard-of-care Prosthetic Foot of One Category Greater Stiffness | Dual Keel Prosthetic Foot | Powered Ankle-foot
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 7
Newtons*seconds/kg
  Walking with no added load | 5.24 (.14) | 5.30 (.14) | 5.27 (.14) | 5.33 (.14) | 5.46 (.15)
  Walking with posterior load | 5.37 (.14) | 5.40 (.14) | 5.42 (.14) | 5.39 (.14) | 5.63 (.15)
  Walking with anterior load | 5.24 (.14) | 5.26 (.14) | 5.29 (.14) | 5.28 (.14) | 5.44 (.15)
  Walking with load on prosthetic side | 5.29 (.14) | 5.29 (.14) | 5.24 (.14) | 5.34 (.14) | 5.51 (.15)
  Walking with load on intact side | 5.25 (.14) | 5.24 (.14) | 5.14 (.14) | 5.21 (.14) | 5.35 (.15)
Statistical Analysis 1: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; Walking with no added load: Hypothesis testing for the overall association between outcome and foot type was carried out using conditional F-tests for each load type; Test type: Superiority; p = 0.100, Regression, Linear
Statistical Analysis 2: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; Walking with posterior load: Hypothesis testing for the overall association between outcome and foot type was carried out using conditional F-tests for each load type; Test type: Superiority; p = 0.032, Regression, Linear
Statistical Analysis 3: Comparison: Standard-of-care Prosthetic Foot vs Powered Ankle-foot; Walking with posterior load: Hypothesis testing for pairwise differences across feet was carried out using Tukey's method to account for the inflation of the Type 1 error due to assessment of 10 pairwise differences for each load; Test type: Superiority; p = 0.024, Regression, Linear
Statistical Analysis 4: Comparison: Dual Keel Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = .046, Regression, Linear
Statistical Analysis 5: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; Walking with anterior load: Hypothesis testing for the overall association between outcome and foot type was carried out using conditional F-tests for each load type; Test type: Superiority; p = .180, Regression, Linear
Statistical Analysis 6: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; Walking with prosthetic side load: Hypothesis testing for the overall association between outcome and foot type was carried out using conditional F-tests for each load type; Test type: Superiority; p = .076, Regression, Linear
Statistical Analysis 7: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; Walking with intact side load: Hypothesis testing for the overall association between outcome and foot type was carried out using conditional F-tests for each load type; Test type: Superiority; p = 0.210, Regression, Linear

2. Primary Outcome: Anterior Ground Reaction Force Impulse (Normalized)
Description: A measure of body forward propulsion. Normalized by body mass, including the mass of the load when applicable.
Time Frame: During study visit (approximately 3 hours)
Measure: Mean (Standard Error); unit: Newtons*seconds/kg
Arm/Group | Standard-of-care Prosthetic Foot | Standard-of-care Prosthetic Foot With Heel-stiffening Wedge | Standard-of-care Prosthetic Foot of One Category Greater Stiffness | Dual Keel Prosthetic Foot | Powered Ankle-foot
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 7
Newtons*seconds/kg
  Walking with no added load | 0.232 (.014) | 0.228 (.014) | 0.213 (.014) | 0.214 (.014) | .257 (.017)
  Walking with posterior load | 0.236 (.014) | 0.236 (.014) | 0.219 (.014) | .225 (.014) | 0.257 (.018)
  Walking with anterior load | 0.225 (.014) | 0.235 (0.014) | 0.212 (.014) | 0.217 (.014) | 0.248 (.017)
  Walking with prosthetic side load | 0.219 (.014) | 0.223 (.014) | 0.213 (.014) | 0.214 (0.014) | 0.256 (.018)
  Walking with intact side load | 0.224 (.014) | 0.219 (0.014) | 0.210 (.014) | 0.208 (0.014) | 0.247 (.014)
Statistical Analysis 1: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.011, Regression, Linear
Statistical Analysis 2: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness; Walking with no added load: Hypothesis testing for pairwise differences across feet was carried out using Tukey's method to account for the inflation of the Type 1 error due to multiple testing; Test type: Superiority; p = .048, Regression, Linear
Statistical Analysis 3: Comparison: Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Powered Ankle-foot; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = .027, Regression, Linear
Statistical Analysis 4: Comparison: Dual Keel Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = .036, Regression, Linear
Statistical Analysis 5: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.044, Regression, Linear
Statistical Analysis 6: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = 0.020, Regression, Linear
Statistical Analysis 7: Comparison: Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness; Walking with anterior load: Hypothesis testing for pairwise differences across feet was carried out using Tukey's method to account for the inflation of the Type 1 error due to multiple testing; Test type: Superiority; p = 0.0085, Regression, Linear
Statistical Analysis 8: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 1, analysis 6]; Test type: Superiority; p = 0.062, Regression, Linear
Statistical Analysis 9: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.045, Regression, Linear

3. Primary Outcome: Peak-to-peak Range of Sagittal Plane Whole-body Angular Momentum (Normalized)
Description: A measure of balance control primarily for anterior and posterior added load conditions. Normalized by body mass (kg) including the mass of the load when applicable, body height (m), and [gravity*body height]^0.5 (m/s) resulting in a unitless number.
Time Frame: During study visit (approximately 3 hours)
Measure: Mean (Standard Error); unit: unitless
Arm/Group | Standard-of-care Prosthetic Foot | Standard-of-care Prosthetic Foot With Heel-stiffening Wedge | Standard-of-care Prosthetic Foot of One Category Greater Stiffness | Dual Keel Prosthetic Foot | Powered Ankle-foot
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 7
unitless
  Walking with no added load | .0172 (.0007) | .0165 (.0007) | .0164 (.0007) | .0160 (.0007) | .0153 (.0007)
  Walking with load on posterior side | .0151 (.0007) | .0150 (.0007) | .0148 (.0007) | .0149 (.0007) | .0145 (.0007)
  Walking with load on anterior side | .0147 (.0007) | .0146 (.0007) | .0147 (.0007) | .0144 (.0007) | .0143 (.0007)
  Walking with load on prosthetic side | .0148 (.0007) | .0144 (.0007) | .0140 (.0007) | .0139 (.0007) | .0138 (.0007)
  Walking with load on intact side | .0144 (.0007) | .0148 (.0007) | .0144 (.0007) | .0145 (.0007) | .0139 (.0007)
Statistical Analysis 1: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; Walking with no load: Hypothesis testing for the overall association between outcome and foot type was carried out using conditional F-tests for each load type; Test type: Superiority; p < 0.010, Regression, Linear
Statistical Analysis 2: Comparison: Standard-of-care Prosthetic Foot vs Dual Keel Prosthetic Foot; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = .0075, Regression, Linear
Statistical Analysis 3: Comparison: Standard-of-care Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = .00007, Regression, Linear
Statistical Analysis 4: Comparison: Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Powered Ankle-foot; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = .032, Regression, Linear
Statistical Analysis 5: Comparison: Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Powered Ankle-foot; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = .044, Regression, Linear
Statistical Analysis 6: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .690, Regression, Linear
Statistical Analysis 7: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 1, analysis 6]; Test type: Superiority; p = .036, Regression, Linear
Statistical Analysis 8: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.400, Regression, Linear

4. Primary Outcome: Peak-to-peak Range of Coronal Plane Whole-body Angular Momentum (Normalized)
Description: A measure of balance control primarily for intact-side added load conditions. Normalized by body mass (kg) including the mass of the load when applicable, body height (m), and [gravity*body height]^0.5 (m/s) resulting in a unitless number.
Time Frame: During study visit (approximately 3 hours)
Measure: Mean (Standard Error); unit: unitless
Arm/Group | Standard-of-care Prosthetic Foot | Standard-of-care Prosthetic Foot With Heel-stiffening Wedge | Standard-of-care Prosthetic Foot of One Category Greater Stiffness | Dual Keel Prosthetic Foot | Powered Ankle-foot
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 7
unitless
  Walking with no added load | 0.0109 (.0009) | .0109 (.0009) | .0111 (.0009) | .0109 (.0009) | .0120 (.0010)
  Walking with load on posterior side | .0094 (.0009) | .0091 (.0009) | .0104 (.0009) | .0100 (.0009) | .0105 (.0010)
  Walking with load on anterior side | .0097 (.0009) | .0096 (.0009) | .0106 (.0009) | .0099 (.0009) | .0113 (.0010)
  Walking with load on prosthetic side | .0103 (.0009) | .0100 (.0009) | .0101 (.0009) | .0103 (.0009) | .0109 (.0010)
  Walking with load on intact side | .0104 (.0009) | .0102 (.0009) | .0106 (.0009) | .0108 (.0009) | .0114 (.0010)
Statistical Analysis 1: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = .079, Regression, Linear
Statistical Analysis 2: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.010, Regression, Linear
Statistical Analysis 3: Comparison: Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness; Walking with posterior load: Hypothesis testing for pairwise differences across feet was carried out using Tukey's method to account for the inflation of the Type 1 error due to multiple testing; Test type: Superiority; p = 0.012, Regression, Linear
Statistical Analysis 4: Comparison: Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Powered Ankle-foot; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = .028, Regression, Linear
Statistical Analysis 5: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p < 0.010, Regression, Linear
Statistical Analysis 6: Comparison: Standard-of-care Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; p = .0094, Regression, Linear
Statistical Analysis 7: Comparison: Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Powered Ankle-foot; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; p = .0025, Regression, Linear
Statistical Analysis 8: Comparison: Dual Keel Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; p = .018, Regression, Linear
Statistical Analysis 9: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 1, analysis 6]; Test type: Superiority; p = .300, Regression, Linear
Statistical Analysis 10: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = .130, Regression, Linear

5. Primary Outcome: Net Positive Ankle Joint Mechanical Work Over the Prosthetic Limb Gait Cycle (Normalized)
Description: Positive ankle joint mechanical work over the prosthetic limb gait cycle is a measure of propulsion capability. A prosthetic foot with greater propulsion capability may enhance gait efficiency during everyday ambulation. Normalized to body mass and the added load mass when applicable.
Time Frame: During study visit (approximately 3 hours)
Measure: Mean (Standard Error); unit: J/kg
Arm/Group | Standard-of-care Prosthetic Foot | Standard-of-care Prosthetic Foot With Heel-stiffening Wedge | Standard-of-care Prosthetic Foot of One Category Greater Stiffness | Dual Keel Prosthetic Foot | Powered Ankle-foot
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 7
J/kg
  Walking with no added load | .158 (.010) | .150 (.010) | .133 (.010) | .127 (.010) | .228 (.025)
  Walking with load on anterior side | .161 (.010) | .161 (.010) | .136 (.010) | .123 (.010) | .231 (.025)
  Walking with load on posterior side | .146 (.010) | .145 (.010) | .124 (.010) | .121 (.010) | .241 (.025)
  Walking with load on intact side | .152 (.010) | .148 (.010) | .126 (.010) | .125 (.010) | .244 (.025)
  Walking with load on prosthetic side | .158 (.010) | .159 (.010) | .136 (.010) | .126 (.010) | .238 (.025)
Statistical Analysis 1: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; Walking with no added load: Hypothesis testing for the overall association between foot and outcome variables was performed using conditional F-tests for each load; Test type: Superiority; p = .0033, Regression, Linear
Statistical Analysis 2: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness; Walking with no added load: Hypothesis testing for pairwise differences across feet was performed using Tukey method to account for the inflation of the Type-1 error due to multiple testing; Test type: Superiority; p = .0001, Regression, Linear
Statistical Analysis 3: Comparison: Standard-of-care Prosthetic Foot vs Dual Keel Prosthetic Foot; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p < 0.0001, Regression, Linear
Statistical Analysis 4: Comparison: Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = .012, Regression, Linear
Statistical Analysis 5: Comparison: Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Dual Keel Prosthetic Foot; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = .0036, Regression, Linear
Statistical Analysis 6: Comparison: Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Powered Ankle-foot; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = .03, Regression, Linear
Statistical Analysis 7: Comparison: Dual Keel Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = .022, Regression, Linear
Statistical Analysis 8: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; Walking with anterior load: Hypothesis testing for the overall association between foot and outcome variables was performed using conditional F-tests for each load; Test type: Superiority; p = 0.0009, Regression, Linear
Statistical Analysis 9: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness; Walking with anterior load: Hypothesis testing for pairwise differences across feet was performed using Tukey method to account for the inflation of the Type-1 error due to multiple testing; Test type: Superiority; p < 0.0001, Regression, Linear
Statistical Analysis 10: Comparison: Standard-of-care Prosthetic Foot vs Dual Keel Prosthetic Foot; [analysis description as in outcome 5, analysis 9]; Test type: Superiority; p < 0.0001, Regression, Linear
Statistical Analysis 11: Comparison: Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness; [analysis description as in outcome 5, analysis 9]; Test type: Superiority; p < 0.0001, Regression, Linear
Statistical Analysis 12: Comparison: Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Dual Keel Prosthetic Foot; [analysis description as in outcome 5, analysis 9]; Test type: Superiority; p < 0.0001, Regression, Linear
Statistical Analysis 13: Comparison: Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Powered Ankle-foot; [analysis description as in outcome 5, analysis 9]; Test type: Superiority; p = 0.03, Regression, Linear
Statistical Analysis 14: Comparison: Dual Keel Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 5, analysis 9]; Test type: Superiority; p = 0.015, Regression, Linear
Statistical Analysis 15: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; Walking with posterior load: Hypothesis testing for the overall association between foot and outcome variables was performed using conditional F-tests for each load; Test type: Superiority; p = 0.0021, Regression, Linear
Statistical Analysis 16: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness; Walking with posterior load: Hypothesis testing for pairwise differences across feet was performed using Tukey method to account for the inflation of the Type-1 error due to multiple testing; Test type: Superiority; p = 0.0002, Regression, Linear
Statistical Analysis 17: Comparison: Standard-of-care Prosthetic Foot vs Dual Keel Prosthetic Foot; [analysis description as in outcome 5, analysis 16]; Test type: Superiority; p = 0.0018, Regression, Linear
Statistical Analysis 18: Comparison: Standard-of-care Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 5, analysis 16]; Test type: Superiority; p = 0.03, Regression, Linear
Statistical Analysis 19: Comparison: Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness; [analysis description as in outcome 5, analysis 16]; Test type: Superiority; p = 0.0004, Regression, Linear
Statistical Analysis 20: Comparison: Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Dual Keel Prosthetic Foot; [analysis description as in outcome 5, analysis 16]; Test type: Superiority; p = 0.0026, Regression, Linear
Statistical Analysis 21: Comparison: Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Powered Ankle-foot; [analysis description as in outcome 5, analysis 16]; Test type: Superiority; p = 0.028, Regression, Linear
Statistical Analysis 22: Comparison: Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Powered Ankle-foot; [analysis description as in outcome 5, analysis 16]; Test type: Superiority; p = 0.0099, Regression, Linear
Statistical Analysis 23: Comparison: Dual Keel Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 5, analysis 16]; Test type: Superiority; p = 0.0085, Regression, Linear
Statistical Analysis 24: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; Walking with intact side load: Hypothesis testing for the overall association between foot and outcome variables was performed using conditional F-tests for each load; Test type: Superiority; p = 0.0021, Regression, Linear
Statistical Analysis 25: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness; Walking with intact side load: Hypothesis testing for pairwise differences across feet was performed using Tukey method to account for the inflation of the Type-1 error due to multiple testing; Test type: Superiority; p < 0.0001, Regression, Linear
Statistical Analysis 26: Comparison: Standard-of-care Prosthetic Foot vs Dual Keel Prosthetic Foot; [analysis description as in outcome 5, analysis 25]; Test type: Superiority; p = 0.0003, Regression, Linear
Statistical Analysis 27: Comparison: Standard-of-care Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 5, analysis 25]; Test type: Superiority; p = 0.033, Regression, Linear
Statistical Analysis 28: Comparison: Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness; [analysis description as in outcome 5, analysis 25]; Test type: Superiority; p = 0.0018, Regression, Linear
Statistical Analysis 29: Comparison: Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Dual Keel Prosthetic Foot; [analysis description as in outcome 5, analysis 25]; Test type: Superiority; p = 0.0043, Regression, Linear
Statistical Analysis 30: Comparison: Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Powered Ankle-foot; [analysis description as in outcome 5, analysis 25]; Test type: Superiority; p = 0.027, Regression, Linear
Statistical Analysis 31: Comparison: Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Powered Ankle-foot; [analysis description as in outcome 5, analysis 25]; Test type: Superiority; p = 0.0095, Regression, Linear
Statistical Analysis 32: Comparison: Dual Keel Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 5, analysis 25]; Test type: Superiority; p = 0.0086, Regression, Linear
Statistical Analysis 33: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Dual Keel Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 5, analysis 24]; Test type: Superiority; p = 0.0016, Regression, Linear
Statistical Analysis 34: Comparison: Standard-of-care Prosthetic Foot vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness; [analysis description as in outcome 5, analysis 25]; Test type: Superiority; p = 0.0007, Regression, Linear
Statistical Analysis 35: Comparison: Standard-of-care Prosthetic Foot vs Dual Keel Prosthetic Foot; [analysis description as in outcome 5, analysis 25]; Test type: Superiority; p < 0.0001, Regression, Linear
Statistical Analysis 36: Comparison: Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Standard-of-care Prosthetic Foot of One Category Greater Stiffness; [analysis description as in outcome 5, analysis 25]; Test type: Superiority; p = 0.0004, Regression, Linear
Statistical Analysis 37: Comparison: Standard-of-care Prosthetic Foot With Heel-stiffening Wedge vs Dual Keel Prosthetic Foot; [analysis description as in outcome 5, analysis 25]; Test type: Superiority; p < 0.0001, Regression, Linear
Statistical Analysis 38: Comparison: Standard-of-care Prosthetic Foot of One Category Greater Stiffness vs Powered Ankle-foot; [analysis description as in outcome 5, analysis 25]; Test type: Superiority; p = 0.02, Regression, Linear
Statistical Analysis 39: Comparison: Dual Keel Prosthetic Foot vs Powered Ankle-foot; [analysis description as in outcome 5, analysis 25]; Test type: Superiority; p = 0.012, Regression, Linear

ADVERSE EVENTS:
Time Frame: 1 week
Description: In this study, subjects only wore the study prosthetic feet while in the laboratory under supervision of laboratory staff. Because the study prosthetic feet could be quickly changed in between walking conditions (no added load, load added to the anterior side, load added to the posterior side, load added to the prosthetic side, and load added to the intact side), adverse events for all arms/groups and interventions were combined.
Arm/Group | Individuals With Lower Limb Amputation
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT07159490/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT07159490/SAP_001.pdf
  • Informed Consent Form (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/90/NCT07159490/ICF_003.pdf